CLINICAL TRIAL: NCT02962167
Title: A Phase 1 Study of Modified Measles Virus (MV-NIS) for the Treatment of Children and Young Adults With Recurrent Medulloblastoma or Recurrent Atypical Teratoid Rhabdoid Tumors (ATRT)
Brief Title: Modified Measles Virus (MV-NIS) for Children and Young Adults With Recurrent Medulloblastoma or Recurrent ATRT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sabine Mueller, MD, PhD (Other)
Collaborators: No More Kids With Cancer (Unknown); The Matthew Larson Foundation for Pediatric Brain Tumors (Other); Vyriad, Inc. (Industry); Mayo Clinic (Other)
Responsible Party: Sponsor-Investigator, Sabine Mueller, MD, PhD, Associate Adjunct Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PNOC 005; 150812 (Other: University of California, San Francisco); NCI-2017-01831 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2016-11-02; First posted 2016-11-11 (Estimated); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Medulloblastoma, Childhood, Recurrent; Atypical Teratoid/Rhabdoid Tumor; Medulloblastoma Recurrent
Keywords: measles virus; recurrent medulloblastoma; recurrent ATRT
MeSH Terms: conditions — Medulloblastoma; Recurrence; Rhabdoid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Locally Recurrent Medulloblastoma/ATRT (Experimental): Patients must have local recurrent disease (defined as negative spine MRI and negative cytology within 21 days prior to study registration) and undergo resection of local recurrence as part of their standard of care. Patients must have undergone what is considered the standard of care as upfront therapy including either surgery followed by high dose chemotherapy with stem cell rescue or multi-modality therapy of surgery, radiation and chemotherapy. Patients will receive the modified measles virus, MV-NIS, directly into the tumor bed during standard of care resection.
  Interventions: Biological: Modified Measles Virus
- Disseminated Recurrent MB/ATRT (Experimental): Patients must have disseminated recurrent medulloblastoma (MB) or ATRT (defined as multifocal disease, positive spine MRI including leptomeningeal disease and/or positive cytology within 21 days prior to study registration) and have adequate CSF flow based on spine MRI with no evidence of bulky disease or if bulky disease is present based on a CSF flow study per institutional guidelines. Patients must have undergone what is considered the standard of care as upfront therapy including either surgery followed by high dose chemotherapy with stem cell rescue or multi-modality therapy of surgery, radiation and chemotherapy. Patients will receive the modified measles virus, MV-NIS, via lumbar puncture (modified measles virus lumbar puncture).
  Interventions: Biological: Modified Measles Virus Lumbar Puncture
- Disseminated Recurrent Medulloblastoma (Experimental): Patients must have disseminated recurrent medulloblastoma (defined as multifocal disease, positive spine MRI including leptomeningeal disease and/or positive cytology within 21 days prior to study registration) and have adequate CSF flow based on spine MRI with no evidence of bulky disease or if bulky disease is present based on a CSF flow study per institutional guidelines. Patients must have undergone what is considered the standard of care as upfront therapy including either surgery followed by high dose chemotherapy with stem cell rescue or multi-modality therapy of surgery, radiation and chemotherapy. Patients will receive the modified measles virus, MV-NIS, via lumbar puncture (modified measles virus lumbar puncture).
  Interventions: Biological: Modified Measles Virus Lumbar Puncture

INTERVENTIONS:
Biological: Modified Measles Virus — Administration of MV-NIS either into the tumor bed, if surgery to remove local tumor
  Other Names: MV-NIS
  Arms: Locally Recurrent Medulloblastoma/ATRT
Biological: Modified Measles Virus Lumbar Puncture — Administration of MV-NIS into the cerebrospinal fluid via lumbar puncture
  Other Names: MV-NIS LP
  Arms: Disseminated Recurrent MB/ATRT; Disseminated Recurrent Medulloblastoma

SUMMARY:
This is a three arm Phase I study within the Pacific Pediatric Neuro-Oncology Consortium (PNOC).

This study will look to determine the safety and recommended phase 2 dose of the modified measles virus (MV-NIS) in children and young adults with recurrent medulloblastoma or atypical teratoid rhabdoid tumor (ATRT).

DETAILED DESCRIPTION:
This is an open label, multi-center, Phase I study to assess the safety of administering MV-NIS directly into the tumor bed (for locally recurrent medulloblastoma or ATRT patients) or into the subarachnoid space (for disseminated recurrent medulloblastoma or ATRT patients).

For locally recurrent patients (patients in the first arm) MV-NIS will be directly administered into the tumor bed following a standard of care surgical resection. For patients with disseminated recurrence (patients in the second or third arm), MV-NIS will be injected via lumbar puncture (LP).

Patients in the second arm will receive a one-time administration of MV-NIS. Patients will be closely monitored for 30 days after injection, and then followed for evaluation of 6 month progressive free survival and overall response rate.

Patients in the third arm will receive two administrations of MV-NIS. Patients will be closely monitored for 56 days after injection, and then followed for evaluation of 4 month progressive free survival.

ELIGIBILITY:
Inclusion Criteria:

• For stratum A, patients must have local recurrent disease (defined as negative spine MRI and negative cytology within 21 days prior to study registration) and undergo resection of local recurrence as part of their standard of care. Children must have undergone what is considered the standard of care as upfront therapy including either surgery followed by high dose chemotherapy with stem cell rescue or multi-modality therapy of surgery, radiation and chemotherapy.

* For stratum B, patients must have disseminated recurrent disease (defined as multifocal disease, positive spine MRI including leptomeningeal disease and/or positive cytology within 21 days prior to study registration) and have adequate cerebrospinal fluid (CSF) flow based on spine MRI with no evidence of bulky disease or if bulky disease is present based on a CSF flow study per institutional guidelines. Children must have undergone what is considered the standard of care as upfront therapy including either surgery followed by high dose chemotherapy with stem cell rescue or multi-modality therapy of surgery, radiation and chemotherapy.
* For stratum C, patients must have disseminated recurrent disease (defined as multifocal disease, positive spine MRI including leptomeningeal disease and/or positive cytology within 21 days prior to study registration) and have adequate cerebrospinal fluid (CSF) flow based on spine MRI with no evidence of bulky disease or if bulky disease is present based on a CSF flow study per institutional guidelines. Children must have undergone what is considered the standard of care as upfront therapy including either surgery followed by high dose chemotherapy with stem cell rescue or multi-modality therapy of surgery, radiation and chemotherapy.

Prior Therapy:

* The patient must have failed at least one prior therapy - surgery followed by high dose chemotherapy with stem cell rescue or multi-modality therapy of surgery, radiation and chemotherapy - prior to study registration. Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study.

  o Myelosuppressive chemotherapy: Patients must have received their last dose of known myelosuppressive anticancer chemotherapy at least three weeks prior to study registration or at least six weeks prior if nitrosourea.

  o Biologic agent: Patient must have recovered from any acute toxicity potentially related to the agent and received their last dose of the biologic agent ≥ 7 days prior to study registration.
* For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended to beyond the time during which adverse events are known to occur. The duration of this interval should be discussed with the study chair.
* For biologic agents that have a prolonged half-life, the appropriate interval since last treatment should be discussed with the Study Chair prior to registration.

  * Monoclonal antibody treatment: At least three half-lives must have elapsed prior to registration. Such patients should be discussed with the study chair prior to registration. For bevacizumab, patients must have received last dose ≥ 32 days prior to study registration.
  * Bone Marrow Transplant: Patient must be:
* ≥ 6 months since allogeneic bone marrow transplant prior to registration
* ≥ 3 months since autologous bone marrow/stem cell prior to registration
* Radiation:

Patients must have:

* Had their last fraction of local irradiation to primary tumor ≥2 weeks prior to registration for local palliative radiation therapy (XRT) (small port)
* Had their last fraction of craniospinal irradiation ≥ 12 weeks prior to registration

  • Age ≥ 12 months to less than or equal to 39 years of age

  • Karnofsky ≥ 50 for patients ≥ 16 years of age, and Lansky ≥ 50 for patients < 16 years of age (See Appendix A). Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score. Patients with pre-existing neurological deficits need to be stable prior to surgery or LP as determined by the investigator.

  • Cluster of Differentiation 4 (CD4) (>= 200/microliter)

  • Organ Function Requirements (within 7 days prior to study registration)
* Adequate Bone Marrow Function Defined as:

  - Peripheral absolute neutrophil count (ANC) ≥ 1000/mm3 and

  - Platelet count ≥ 100,000/mm3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment).
* Adequate Renal Function Defined as:

  * Creatinine clearance or radioisotope glomerular filtration rate (GFR) greater than or equal to 70 milliliters (mL)/min/1.73 m2 or
  * A serum creatinine based on age/gender as follows:

Maximum Serum/Creatinine (mg/dL)

Age Male Female

1. - 2 years 0.6 0.6
2. to <6 years 0.8 0.8

6 to <10 years 1 1

10 to <13 years1.2 1.2

13 to <16 years1.5 1.4

* 16 years 1.7 1.4 The threshold creatinine values in this table were derived from the Schwartz formula for estimating GFR utilizing child length and stature data published by the Centers for Disease Control and Prevention (CDC).

  * Adequate Liver Function Defined as:

    - Bilirubin (sum of conjugated + unconjugated) less than or equal to 1.5 x upper limit of normal (ULN) for age and

    - serum glutamic-pyruvic transaminase (SGPT)/alanine aminotransferase (ALT) less than or equal to 110 U/L and

    - Serum albumin less than or equal to 2 g/dL.

    • The effects of MV-NIS on the developing human fetus are unknown. For this reason, females of child-bearing potential and males must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and 4 months after completion of MV-NIS administration. Should a female become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

    • Ability to understand and the willingness to sign a written informed consent document.

    -Exclusion Criteria

    -Patients who have had chemotherapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C) or radiotherapy within 2 weeks prior to entering the study for local palliative XRT (small port) and within 12 weeks prior for patients that received craniospinal XRT

    - Patients who have not recovered from acute adverse events due to agents administered more than 4 weeks earlier

    -Patients who are receiving any other investigational agents

    - History of allergic reactions attributed to compounds of similar chemical or biologic composition to measles virus vaccination

    -Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

    -Female patients of childbearing potential must not be pregnant or breast-feeding.

    -Female patients of childbearing potential must have a negative serum or urine pregnancy test (within 7 days prior to study registration)

    -Patients with known HIV positivity
    * Patients with inability to return for follow-up visits or obtain follow-up studies required to assess toxicity to therapy
    * Exposure to household contact with known immunodeficiency
    * History of chronic hepatitis B or C infection
    * History of organ transplantation
    * Patients with evidence of extraneural disease
    * Patients on chronic steroids or other immunosuppressive agents. Note: Patients that are currently using inhaled, intranasal, ocular, topical or other non-oral or non-IV steroids may be eligible.
    * Inability to undergo magnetic resonance (MR) imaging to assess disease status

Ages: 12 Months to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-05-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as Assessed by CTCAE v5. | 12 months
  The safety of the modified measles virus will be assessed by monitoring for adverse events. Subjects will be monitored for adverse events via scheduled laboratory assessments, vital sign measurements, and physical examinations. The severity of any toxicity will be graded according to the NCI CTCAE v5.0. We will aggregate this information into the number of subjects with adverse events that are related to study treatment.
Recommended Phase 2 Dose. | 12 months
  The maximum tolerated dose (MTD)/recommended phase 2 dose (RP2D) will be the dose level at which 6 evaluable patients have been treated and at most 1 patient experienced a dose limiting toxicity (DLT) and the next highest dose level is too toxic or we have reached the protocol defined highest dose level.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 24 months
  Any eligible patient that receives MV-NIS will be considered evaluable for clinical efficacy. The objective response criteria is that partial response (PR) and complete response (CR) must be confirmed at least 8 weeks after the initial PR or CR criteria is met.
Progression Free Survival (PFS) | 24 months
  For patients who are still progression free at the time of analysis, PFS will be censored at the last contact date. PFS will be estimated using the Kaplan-Meier method.

OTHER OUTCOMES:
The distribution of MV-NIS | 12 months
  Subjects who consent to this optional study will receive an injection of technetium-99m (TC-99m) (pertechnetate) and then undergo SPECT imaging to determine MV-NIS distribution after local injection or after administration into the subarachnoid space.

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Mueller, MD, PhD, MAS, Study Chair — University of California, San Francisco
Locations (8):
- United States (8):
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Washington University in St. Louis, St Louis, Missouri
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No